CLINICAL TRIAL: NCT01177917
Title: Evaluation of Mineral Absorption in Infants Fed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Other Study IDs: 3371-4
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Mineral Absorption in the Urine
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cow milk-based infant formula with prebiotic blend (Experimental)
  Interventions: Other: Infant Formula
- Marketed Cow milk-based infant formula (Placebo Comparator)
  Interventions: Other: Infant Formula

INTERVENTIONS:
Other: Infant Formula

SUMMARY:
This clinical trial will help determine if prebiotics can increase mineral absorption in babies

ELIGIBILITY:
Inclusion Criteria:

* Singleton
* Term infant
* Birth weight of 2500 g or more
* 56-70 days of age
* Signed informed consent
* Consuming a cow's milk-based infant formula for at least 24 hours.

Exclusion Criteria:

* History of underlying disease or congenital malformation which, in the opinion of the Investigator, is likely to interfere with the normal growth and development or the evaluation of the mineral absorption of the participant
* Use of multiple vitamin and mineral supplements prior to enrollment.
* Evidence of formula intolerance or poor intake at time of randomization

Ages: 56 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the amount of minerals in the urine

SECONDARY OUTCOMES:
Compare the amount of vitamins and minerals in the blood

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Children's Hospital of Iowa, Coralville, Iowa
  - Pediatric Clinical Trials Unit, Louisville, Kentucky
  - The Center for Human Nutrition, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center Clinical Trials Office, Cincinnati, Ohio
  - Children's Research and Nutrition Center, Houston, Texas